CLINICAL TRIAL: NCT07315009
Title: An Active Fundament, Fundamentally Better: From an Early Age, Moving Well and Moving Enough as the Basis for a Lifetime of Physical Activity.
Brief Title: Active Fundament - Fundamentally Better
Acronym: AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fontys University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Jasper de Graef, Teacher-researcher (PhD Candidate), Fontys University of Applied Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FHML-REC/2024/032; RAAK.PRO05.034 (Other Grant/Funding Number: Nation agency of applied research (Regieorgaan SIA))
Record Dates: First submitted 2025-12-04; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Physical Inactivity in Early Childhood and Care; Delayed Fundamental Motor Skill Development; Early Childhood & Care Physical Activity Behavior; Motor Development in Children Aged 2-6 Years; Physical Activity-Supportive Early Childhood Education and Care (ECEC) Environment
Keywords: Child center; physical activity levels; preschool; childcare; motor skills

STUDY DESIGN:
Intervention Model Description: Longitudinal, Quasi-experimental.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Childeren in ECEC settings (Experimental): 2-6 year olds
  Interventions: Behavioral: Actief Fundament
- Professionals in ECEC settings (Experimental): Pedagogical and educational staff including management
  Interventions: Behavioral: Actief Fundament

INTERVENTIONS:
Behavioral: Actief Fundament — In procesmeetings with the intervention centers we will discuss possible changes to improve physical activity levels of children. Activities and changes will be based on the measurement outcomes.

SUMMARY:
The objective of this longitudinal, quasi-experimental study is to improve children's fundamental motor skills and physical activity levels. In addition, the study aims to support pedagogical staff and educators in implementing physical activity during the workday, with the intention of facilitating a more supportive and enjoyable working environment that aligns with children's needs for physical activity.

The study is conducted in 18 child centers, combining childcare and preschool settings. Participants include children aged 2-6 years and their pedagogical staff and teachers.

The primary research questions addressed are:

* Can pedagogical staff and teachers be supported in increasing physical activity levels among children aged 2-6 years?
* Can a scalable intervention for child centers be developed that can be implemented in other regions following completion of the study? A total of nine intervention centers will be compared with nine control centers to determine whether observed effects can be attributed to the intervention.

Children will participate in assessments of motor skills, wear accelerometers to measure physical activity levels, and take part in walk-along interviews and a draw-and-tell method. Parents will complete questionnaires. Pedagogical staff and teachers will complete questionnaires and participate in observational assessments. Management representatives of the child centers (both preschool and childcare) will participate in interviews and complete a questionnaire to construct an echogram.

ELIGIBILITY:
Inclusion Criteria:

* Children must be in the child center in the recruitment period(s)
* Professionals in ECEC and management must be working at the child center during the recruitment period.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Average daily light physical activity, moderate-to-vigorous physical activity (MVPA), and sedentary behavior in minutes, assessed by accelerometry | One week of accelerometer measurement, repeated annually in the spring season for four consecutive years
  Children's physical activity behavior will be objectively assessed using triaxial accelerometers (ActiGraph GT3X+). Accelerometers will be worn during waking hours for seven consecutive days. Physical activity data will be processed using validated pediatric cut-points to derive average daily time spent in light physical activity, moderate-to-vigorous physical activity (MVPA), and sedentary behavior. Outcomes will be reported as mean minutes per day for each activity intensity category per measurement period.
Pedagogical support for physical activity assessed by the Movement Environment Rating Scale (MOVERS) | Assessed at baseline, mid-intervention, and at study completion (approximately 3 years)
  Pedagogical actions of teachers and caretakers that support children's physical activity will be assessed using the Movement Environment Rating Scale (MOVERS). MOVERS is an observational instrument designed for early childhood education and care settings and evaluates the extent to which pedagogical practices and environmental characteristics promote physical activity and motor development. The scale consists of four domains and yields a total score ranging from 1 to 7, with higher scores indicating a more supportive physical activity environment and higher-quality pedagogical practices. Observations will be conducted during a full day in childcare and preschool settings by trained observers.
Self-reported pedagogical physical activity practices assessed by questionnaire | Assessed at baseline and annually thereafter during the spring season, through study completion (up to 4 years)
  Pedagogical staff's self-reported practices related to promoting physical activity and fundamental motor skills will be assessed using a structured questionnaire. The questionnaire captures frequency and type of physical activity-related pedagogical actions during the workday. Outcomes will be summarized as mean scores per domain, with higher scores indicating greater engagement in physical activity-supportive practices.

SECONDARY OUTCOMES:
Motor competence assessed by the Athletic Skills Track (AST) | Assessed at baseline and annually thereafter during the spring season, through study completion (up to 4 years)
  Motor competence will be assessed using the Athletic Skills Track (AST), a standardized motor competence assessment for children. The AST consists of a sequence of age-appropriate motor tasks assessing balance, coordination, agility, jumping, and running skills. Performance is expressed as total completion time in seconds, with lower times indicating better motor skill performance. Only children aged 4 years and older will be assessed.
Motor competence assessed by the 4 Skills Scan (4SS) test | Assessed at baseline and annually thereafter during the spring season, through study completion (up to 4 years)
  Motor competence will be assessed using the 4 Skills Scan (4SS) test, a validated motor skill assessment for children. The 4SS evaluates four motor domains: jumping force, jumping coordination, running coordination, and object control. Each domain is scored on a standardized scale, resulting in a total score ranging from 4 to 16, with higher scores indicating better motor skill proficiency. Only children aged 4 years and older will be assessed.
Parental involvement in the child center and child physical activity assessed by questionnaire | Assessed at baseline and annually thereafter during the spring season, through study completion (up to 4 years)
  Parental involvement will be assessed using a structured parent questionnaire. The questionnaire measures parental involvement across multiple domains, including involvement in the child center, support for the child's physical activity, and perceived child well-being. Domain-specific mean scores will be calculated, with higher scores indicating greater parental involvement and support. The questionnaire will be administered to parents of participating children.

CONTACTS AND LOCATIONS:
Overall Officials: Dave van Kann, PhD, Study Director — Fontys University of Applied Sciences; Jessica Gubbels, Associate Professor, Study Director — Maastricht University
Locations (3):
- Netherlands (3):
  - Maastricht University, Maastricht, Limburg
  - Fontys Sport en Bewegen, Eindhoven, North Brabant
  - Hogeschool van Amsterdam, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study project website — http://www.actieffundament.nl
- See also: Project funding — https://www.sia-projecten.nl/project/een-actief-fundament-fundamenteel-beter-van-jongs-af-aan-goed-en-voldoende-bewegen-als-basis-voor-een-leven-lang-bew